CLINICAL TRIAL: NCT01538693
Title: Molecular Markers of Neuroplasticity During High-Intensity Exercise in Subjects With Incomplete Spinal Cord Injury
Brief Title: Molecular Markers of Neuroplasticity During Exercise in People With Incomplete Spinal Cord Injury
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: T. George Hornby (Other)
Collaborators: University of Medicine and Dentistry of New Jersey (Other); Shirley Ryan AbilityLab (Other)
Responsible Party: Sponsor-Investigator, T. George Hornby, Assistant Professor, Shirley Ryan AbilityLab
Organization: Shirley Ryan AbilityLab (Other)
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Basic Science
Other Study IDs: STU00056144
Record Dates: First submitted 2012-01-24; First posted 2012-02-24 (Estimated); Last update posted 2015-05-19 (Estimated); Status verified 2015-05

CONDITIONS: Spinal Cord Injury
Keywords: BDNF; serotonin; high-intensity; exercise
MeSH Terms: conditions — Spinal Cord Injuries; Motor Activity | interventions — Escitalopram; Cyproheptadine; Sugars

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (3):
- escitalopram oxalate (Active Comparator): Exercise testing with escitalopram oxalate dose
  Interventions: Drug: escitalopram oxalate; Other: Graded intensity exercise
- cyproheptadine (Active Comparator): exercise testing with cyproheptadine dose
  Interventions: Drug: Cyproheptadine; Other: Graded intensity exercise
- placebo (Placebo Comparator): exercise testing with placebo dose
  Interventions: Drug: sugar pill; Other: Graded intensity exercise

INTERVENTIONS:
Drug: escitalopram oxalate — 10 mg 4.5 hours prior to testing
  Other Names: Lexapro
  Arms: escitalopram oxalate
Drug: Cyproheptadine — 8mg 4.5 hours prior to testing
  Arms: cyproheptadine
Drug: sugar pill — 4.5 hour prior to testing
  Arms: placebo
Other: Graded intensity exercise — modified bruce protocol for peak oxygen consumption testing

SUMMARY:
The purpose of this study is to determine whether exercising (walking) at different intensities increases levels of factors in the blood and saliva that are known to impact neuroplasticity (how the connections in the spinal cord and brain can change) and if these levels are changed by pairing exercise with a single dose of commonly used prescription drugs or by your mood.

DETAILED DESCRIPTION:
The protein brain-derived neurotrophic factor (BDNF) is known to promote cell survival, improve synaptic function, and induce neuronal morphological changes. Consequently, BDNF plays a major role in neuroplasticity and the ability of the central nervous system to adapt and recover following injury. Regardless of the molecular mechanisms by which this occurs (which are poorly understood), potentiating the expression of BDNF following spinal cord injury has been shown to improve functional outcomes in animals.(1, 2) It is well documented in both animal and human literature that the production BDNF increases with physical exercise in healthy populations and individuals with chronic disease or disability. (3) The literature suggests that this increase is proportional to the intensity of exercise, though the parameters of exercise to maximize this effect are poorly understood. (2, 4-6) From animal research, it has been postulated that serotonin (5HT) plays a role in the mechanism of increase in BDNF expression, (7-9) with findings that specifically demonstrate potentiation of the exercise-induced expression with antidepressant treatment(10)and a blunted response when monoaminergic signaling is blocked.(11) A specific genetic variation in the BDNF gene, found in approximately 30% of the population has also been noted as an important factor in the proper release of BDNF with associated deficits in motor learning. (12, 13) Initial evidence also suggests that this polymorphism may have an impact of the relationship between exercise and BDNF. (14, 15) The objective of this study is the evaluate the response of serum concentrations of brain-derived neurotrophic factor ([BDNF]s) to an acute bout of exercise in ambulatory people with incomplete spinal cord injury; additionally, to examine the effect of pharmacological agents that alter serotonergic (5HT) transmission on this exercise-induced change in [BDNF]s. To achieve this objective we will investigate [BDNF]s during a treadmill test alone and in combination with two commonly used medications; escitalopram oxalate , a selective-5HT reuptake inhibitor (SSRI) and cyproheptadine (CYPRO), a 5HT antagonist.

Studies have also shown a relationship of BDNF to mood, in particular, depression. A secondary study will be performed in parallel with the primary study with the purpose of examining mood and how it correlates with the molecular markers for neuroplasticity as individuals participate in the repeated exercise and the other stated interventions. As the subjects progress over the course of the study time mood may change and may impact the relationship of the BDNF to the primary interventions.

ELIGIBILITY:
Inclusion Criteria:

* Must be motor incomplete spinal cord injury (ASIA C or D) of 1 year or greater duration, with anatomical lesions between C1-T10
* Must be between 18 and 75 years of age
* Must be ambulatory with passive range of motion consistent with normal walking, and must include: ankle dorsiflexion ankle to 10° and plantarflexion to 30°, knee flexion from 0 to 90°, hip flexion/extension to 90° to -10°.
* Must be medically stable with medical clearance to participate, with absence of concurrent severe medical illness including: unhealed decubiti, existing infection, significant cardiovascular or metabolic disease which limits exercise participation, significant osteoporosis (as indicated by history of fractures following injury), active heterotrophic ossification in the lower extremities, known history of peripheral nerve injury in lower legs, history of known traumatic head injury, mental illness, history of pre-existing QT interval prolongation, congenital long QT syndrome, and history of pulmonary complications, including significant obstructive and/or restrictive lung diseases
* May be undergoing concurrent physical therapy
* May be of childbearing potential (for women)
* Men and women will be recruited for participation in the proposed study at rates consistent with national and local average of gender disparities of SCI (80% male, 20% women)
* Individuals of different ethnicities will be recruited at rates similar to the national and local ethnicity rates. Current data since 2005 indicate that of the entire population of SCI, 66.1% are Caucasian, 27.1% are African American, 6.6% are of Hispanic origin, and 2.0% are Asian.

Exclusion Criteria:

* Weighing more than 300lbs
* Ventilator-dependency
* Use of substantial orthopedic bracing to stabilize the cervical or thoracic vertebral column
* Inability to tolerate 10 minutes of standing without orthostasis (decrease in blood pressure by 20 mmHg systolic and 10 mmHg diastolic).
* Women who are pregnant or who are considering becoming pregnant will be excluded due to the trunk and pelvis restraints required for use during locomotion, and secondary to the unknown effects of the pharmacological agents on the developing fetus
* Exhibiting symptoms suggestive of depression according to the Personal health Questionaire (PHQ-9)
* Subjects who exhibit hemoglobin levels consistent with anemia (<13g/dL for men and <12g/dL for women) will be excluded from the study.
* Currently taking prescribed anti-depressant medications, including specific monoaminergic agents, their precursors or their agonists, antipsychotics, medications known to prolong the QT interval, or other medications with known interactions to the SSRIs. All subjects will be excluded from participation unless both attending physician and patient agree to cease all such medications during the evaluation and training period. A 14-day washout period for SSRIs and a 72 hour washout for Tizanidine will be utilized. Subjects will be financially responsible for the physician visits necessary to wean from medication. Completion of appropriate and safe weaning will be confirmed by the patients' physician.
* Currently taking prescribed anti-spastic medications. Specific agents to be excluded include baclofen (Lioresal®) and benzodiazepines (Diazepam®). Selected agents used for pain modulation will be evaluated per subject to ascertain potential interactions with test agent. All subjects will be excluded from participation unless both attending physician and patient agree to cease all such medications during the evaluation and training period. A 72-hour minimum washout period for all such medications will be utilized. Subjects will be financially responsible for the physician visits necessary to wean from medication. Completion of appropriate and safe weaning will be confirmed by the patients' physician.
* Clinically diagnosed liver, renal, or other metabolic disease that may interfere with drug action and/or clearance

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2011-12; Primary Completion 2015-05 (Actual); Study Completion 2015-05 (Actual)

PRIMARY OUTCOMES:
Change in blood serum concentration of neuroplastic proteins | assessed prior to, throughout, and following the duration of a graded exercise test, over an expected average of 2 hours
  During a graded treadmill test, 5mL of blood will be taken at each speed the subject is able to obtain before failure. 5mL of blood will also be taken immediately after completion of the treadmill test and every 10 minutes for up to 30 minutes after completion.

SECONDARY OUTCOMES:
fastest possible walking velocity overground | one time, baseline measure
Six Minute Walk Distance | one time basline measurement
Volitional strength: Lower Extremity Motor Score | one time baseline measure
Modified Ashworth Scale | one time baseline measurement
Spinal Cord Assessment tool for Spasticity | one time baseline measure
Measure of Community mobility | Step activity monitor worn on lower extremity for 7 days
Sagittal plane kinematics of excursions of hip/knee/ankle | continuous assessment for an average of ten minutes at each visit
Peak ambulation velocity | One time measure at the end of each graded intensity treadmilll test
Oxygen consumption | continuous assessment for an average of ten minutes at each visit
Heart Rate | continuous assessment for an average of ten minutes at each visit
Rating of Perceived Exertion (Borg Scale) | continuous assessment for an average of ten minutes at each visit

CONTACTS AND LOCATIONS:
Overall Officials: Thomas G Hornby, PhD, PT, Principal Investigator — University of Illinois at Chicago, Rehabiliation Institute of Chicago, Northwestern University
Locations (1):
- Rehabiliation Institute of Chicago, Chicago, Illinois, United States

REFERENCES:
- [Background] Ying Z, Roy RR, Zhong H, Zdunowski S, Edgerton VR, Gomez-Pinilla F. BDNF-exercise interactions in the recovery of symmetrical stepping after a cervical hemisection in rats. Neuroscience. 2008 Sep 9;155(4):1070-8. doi: 10.1016/j.neuroscience.2008.06.057. Epub 2008 Jul 3. PMID 18672032
- [Background] Ying Z, Roy RR, Edgerton VR, Gomez-Pinilla F. Exercise restores levels of neurotrophins and synaptic plasticity following spinal cord injury. Exp Neurol. 2005 Jun;193(2):411-9. doi: 10.1016/j.expneurol.2005.01.015. PMID 15869943
- [Background] Knaepen K, Goekint M, Heyman EM, Meeusen R. Neuroplasticity - exercise-induced response of peripheral brain-derived neurotrophic factor: a systematic review of experimental studies in human subjects. Sports Med. 2010 Sep 1;40(9):765-801. doi: 10.2165/11534530-000000000-00000. PMID 20726622
- [Background] Ferris LT, Williams JS, Shen CL. The effect of acute exercise on serum brain-derived neurotrophic factor levels and cognitive function. Med Sci Sports Exerc. 2007 Apr;39(4):728-34. doi: 10.1249/mss.0b013e31802f04c7. PMID 17414812
- [Background] Cotman CW, Berchtold NC. Exercise: a behavioral intervention to enhance brain health and plasticity. Trends Neurosci. 2002 Jun;25(6):295-301. doi: 10.1016/s0166-2236(02)02143-4. PMID 12086747
- [Background] Neeper SA, Gomez-Pinilla F, Choi J, Cotman CW. Physical activity increases mRNA for brain-derived neurotrophic factor and nerve growth factor in rat brain. Brain Res. 1996 Jul 8;726(1-2):49-56. PMID 8836544
- [Background] Ivy AS, Rodriguez FG, Garcia C, Chen MJ, Russo-Neustadt AA. Noradrenergic and serotonergic blockade inhibits BDNF mRNA activation following exercise and antidepressant. Pharmacol Biochem Behav. 2003 Apr;75(1):81-8. doi: 10.1016/s0091-3057(03)00044-3. PMID 12759116
- [Background] Nibuya M, Morinobu S, Duman RS. Regulation of BDNF and trkB mRNA in rat brain by chronic electroconvulsive seizure and antidepressant drug treatments. J Neurosci. 1995 Nov;15(11):7539-47. doi: 10.1523/JNEUROSCI.15-11-07539.1995. PMID 7472505
- [Background] Russo-Neustadt AA, Beard RC, Huang YM, Cotman CW. Physical activity and antidepressant treatment potentiate the expression of specific brain-derived neurotrophic factor transcripts in the rat hippocampus. Neuroscience. 2000;101(2):305-12. doi: 10.1016/s0306-4522(00)00349-3. PMID 11074154
- [Background] Russo-Neustadt A, Beard RC, Cotman CW. Exercise, antidepressant medications, and enhanced brain derived neurotrophic factor expression. Neuropsychopharmacology. 1999 Nov;21(5):679-82. doi: 10.1016/S0893-133X(99)00059-7. PMID 10516964
- [Background] Garcia C, Chen MJ, Garza AA, Cotman CW, Russo-Neustadt A. The influence of specific noradrenergic and serotonergic lesions on the expression of hippocampal brain-derived neurotrophic factor transcripts following voluntary physical activity. Neuroscience. 2003;119(3):721-32. doi: 10.1016/s0306-4522(03)00192-1. PMID 12809693
- [Background] Pearson-Fuhrhop KM, Cramer SC. Genetic influences on neural plasticity. PM R. 2010 Dec;2(12 Suppl 2):S227-40. doi: 10.1016/j.pmrj.2010.09.011. PMID 21172685
- [Background] Cheeran B, Talelli P, Mori F, Koch G, Suppa A, Edwards M, Houlden H, Bhatia K, Greenwood R, Rothwell JC. A common polymorphism in the brain-derived neurotrophic factor gene (BDNF) modulates human cortical plasticity and the response to rTMS. J Physiol. 2008 Dec 1;586(23):5717-25. doi: 10.1113/jphysiol.2008.159905. Epub 2008 Oct 9. PMID 18845611
- [Background] Bryan A, Hutchison KE, Seals DR, Allen DL. A transdisciplinary model integrating genetic, physiological, and psychological correlates of voluntary exercise. Health Psychol. 2007 Jan;26(1):30-9. doi: 10.1037/0278-6133.26.1.30. PMID 17209695
- [Background] Mata J, Thompson RJ, Gotlib IH. BDNF genotype moderates the relation between physical activity and depressive symptoms. Health Psychol. 2010 Mar;29(2):130-3. doi: 10.1037/a0017261. PMID 20230085